CLINICAL TRIAL: NCT04214314
Title: Efficacy of a Computerized Program of Cognitive Rehabilitation of Attention in People With Acquired Brain Injury (ABI): Pilot Study
Brief Title: Efficacy of a Computerized Program of Cognitive Rehabilitation of Attention in People With Acquired Brain Injury (ABI)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ikerbasque - Basque Foundation for Science (Other)
Responsible Party: Principal Investigator, Juan Carlos Arango Lasprilla, Neuropsychologist- Researcher, Ikerbasque - Basque Foundation for Science
Other Study IDs: 001b
Record Dates: First submitted 2019-12-22; First posted 2020-01-02 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Brain Injuries
Keywords: Attention; Acquired Brain Injury; Attentional Program; Intervention of attention; Spanish adults; Rehabilitation program
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: The control group will continue to receive the integral rehabilitation provided by the center.
- Experimental: The participants of the experimental group, in addition to the integral rehabilitation of the center will receive the training of the attention through NeuronUp APT. There will be 3 rehabilitation sessions of one hour a week for about a month and a half or two.
  Interventions: Behavioral: NeuronUp APT attentional program

INTERVENTIONS:
Behavioral: NeuronUp APT attentional program — NeuronUp APT attentional program consists of 4 types of attention with 20 activities each and 5 different levels of difficulty per activity. These 20 activities will be divided into two blocks (block A or block B) of 10 activities each and then, randomly, participants will be administered one block or another. The administration of the entire program is approximately one month and a half or 2 months per patient, with sessions of one hour, 3 times per week.
  Groups: Experimental

SUMMARY:
Acquired Brain Injury (ABI) is a sudden lesion in the brain, not congenital or perinatal,caused by various pathologies.According to the National Statistics Institute,in Spain 78% of people suffering from ABI are a result of stroke,and 22% due to Traumatic Brain Injuries (TBIs) and other causes.The ABI is in most cases with problems of cognitive,physical,emotional,social,family and work.Of all these problems,attentional alterations are one of the most frequent and disabling for these participants,with a prevalence of 30-62%.However,there are currently no specific programs for the rehabilitation of attentional processes in people with ABI in Spain.So recently,a program focused on the rehabilitation of NeuronUp APT attentional processes has been developed,based on the theoretical model of Sohlberg and Mateer,which considers attention as a multidimensional cognitive function that is hierarchically organized.This program includes a large group of rehabilitation activities in contexts similar to those of daily life.Objectives:1)Evaluate the effectiveness of the NeuronUp APT attentional training program for the improvement of the attention problems presented by participants with ABI;2)determine whether the improvement of attention problems in participants with ABI causes changes in their functioning emotional and quality of life and 3)determine whether the improvement of the attention problems in participants with ABI causes changes in the functionality of the participants and, consequently, in the activities of their daily lives.Method:This is a randomized clinical trial, 46 participants with ABI between the ages of 18-65 will be recruited; 23 participants will be assigned to the experimental group (integral rehabilitation+NeuronUp APT) and the other 23 to the control group (integral rehabilitation) randomly,using a simple randomization method.Both groups will be evaluated before the start of the intervention, after the end of the intervention and 6 months after the intervention, thus collecting sociodemographic information,clinical characteristics of the disease, cognitive screening measures,emotional functioning test,functional and quality of life.Conclusions:It is hoped to achieve a transfer of the gains obtained,through the training of the attention through the NeuronUp APT rehabilitation program,to other aspects of cognitive,emotional functioning and quality of life.It is also expected that these people improve their attention problems in their daily lives.

DETAILED DESCRIPTION:
General objectives

1)Evaluate the effectiveness of the NeuronUp APT attention training program for the improvement of the attention problems presented by participants with ABI. 2)Determine whether the improvement of the attention problems in the group of participants with ABI, leads to an improvement in the cognitive performance of these participants in the other areas of cognitive functioning. 3)Determine if the improvement of attention problems in participants with ABI, causes changes in their emotional functioning and quality of life. 4)Determine if the improvement of the attention problems in participants with ABI, causes changes in the functionality of the participants and, consequently, in the activities of their daily life.

Specific objectives

1)Determine if there are significant differences between the groups in the scores of the attention tests over time. 2)Determine if there are significant differences between the groups in the scores of the neuropsychological tests that measure memory, executive functions and language over time. 3)Determine if there are significant differences between the groups in the scores of the scale of attention problems in daily life after the intervention.4)Determine if there are significant differences between the groups in the scores of the scale of quality of life over time. 5)Determine if there are significant differences between the groups in the scores of the scales of emotional functioning over time. 6)Determine if there are significant differences between the groups in the scores of the functional functioning scales over time.

Hypothesis

1)Participants in the experimental group will present significantly higher scores in the neuropsychological tests that evaluate the attention at the end of the intervention and six months later compared to the control group. 2)Participants in the experimental group will present significantly higher scores on neuropsychological tests that assess memory, language and executive functions at the end of the intervention and 6 months later compared to the control group. 3)Participants in the experimental group will present significantly lower scores on the scales that measure attention problems in daily life, both at the end of the intervention and at six months later compared to the control group.4)The gains observed in the attentional functioning of the participants of the experimental group will be reflected in an improvement of their emotional functioning, their functional status and their quality of life at the end of the intervention and six months later compared to the control group.

Brief Summary of approach and methodology

- Participants: 46 participants will be recruited with stroke, aged between 18 and 65, who attend the Acquired Brain Injury Unit of the Aita Menni Hospital (Mondragón-Arrasate); specifically, the investigators will focus on participants whose diagnosis is moderate-severe TBI and patients with a diagnosis of stroke, in the last three years. To determine the sample size, a statistical power analysis was carried out with the G *Power program. For this, the Cohen criteria have been taken into account, so that an effect size of 0.45 (large for the ANOVA statistic) and alpha and beta values of 0.05 and 0.95, respectively, have been established. The information will be obtained from each participant at three specific times: before to the start of the intervention, after completing the implementation of the program and six months after the end of the program.

The information that will be collected in each of these three times is as follows:

* Sociodemographic data Information on age, years of schooling (number of years), gender (male vs. female), occupation (employed, unemployed, student, retired, etc.), marital status (single, married, free union) will be collected through the interview, laterality (right-handed, left-handed, ambidextrous) and monthly economic income (total amount of income).
* Clinical characteristics, screening tests: Primary Outcomes Measures.
* Study of cognitive functioning, study of the attentional state in the participant's daily life, study of the emotional state of participants, study of the emotional state of participants,Quality of life study,Study of functional status: Secondary Outcomes Measures.

NeuronUp APT attentional program

The model by which NeuronUp APT is governed is the clinical rehabilitation model described by Sholberg and Mateer, which considers attention as a main cognitive function of a multidimensional character that is hierarchically organized.NeuronUp APT is composed of 80 activities, based on activities of daily living whose objective is to achieve the greatest possible ecology and a true transfer of cognitive training to the daily activities of patients. All activities are computerized and can be performed on any electronic device, computer, mobile and tablet, allowing patients to continue training from home.

Since it is based on the traditional clinical model, program activities are organized according to the type of attention in blocks of 20 exercises, as follows:

* Sustained attention: Exercises in which a series of visual or auditory stimuli are presented to the participant, depending on the activity, of which there is a Target Stimulus (TS). The stimuli appear one by one on the electronic device, and each time the participant sees or hears the TS, the person must press on the screen. For example, in one of the activities the participant is instructed to delete the photos of his/her cat from the mobile. To do this, different photos appear on the screen of a mobile phone, and the participant's task is to press each time the photo of the cat comes out.
* Selective attention: Exercises in which in addition to visual or auditory stimuli other distracting stimuli are presented, such as ambient noise in the case of visual activities, or videos in the case of auditory activities. For example, in one of the activities is simulated that the participant is in a shopping center and must attend to the license plates of the cars that are being announced by public address system because the cars are badly parked. To do this, a video of a shopping center full of people is presented while listening to the auditory stimuli, in this case, the license plates of the cars, and the task of the participant is to press on the screen every time hear a registration ending in a certain number.
* Alternate attention: Exercises in which there are two TSs that alternate. For example, in one of the activities, the participant is told that is at an airport and must collect his/her bags and those of a relative. To do this, the participant must first attend and press each time see a specific suitcase (first TS), and when hears an alarm the participant must change the instruction and press each time see another particular suitcase (second TS).
* Divided attention: Exercises in which a visual and auditory stimulus are simultaneously presented, which the participant must process at the same time. For example, in one of the activities, the participant is instructed to attend the traffic signs and press every time sees the signal that indicates the possible appearance of deer to reduce speed. In addition, the participant must follow the Global Positioning System (GPS) instructions and press each time the instruction indicates the presence of a radar. Since the way to respond to the stimuli is by pressing on the screen, the two TSs are never presented at the same time, since otherwise would not be possible to determine which of the two stimuli the participants are attending.

The difficulty of each of the tasks will be progressively increased, depending on the number of stimuli and the time spent, through 5 levels. So, in the lower levels the tasks last less and contain less stimuli than in the upper ones. Thus, during the training process, patients complete all levels of sustained attention activities, and then start the selective attention block, then the alternate attention, and finally the divided attention. For the implementation of NeuronUp APT, the neuropsychologist will need to make use of a neurorehabilitation web platform.

Statistical analysis by objectives

In the first place, preliminary analyzes will be carried out by means of a t-test to determine if there are differences in the sociodemographic variables between groups (sex, age, schooling).Subsequently, multiple analyzes of 2 X 3 ANOVAS will be carried out, both of repeated measures intra and between groups, where the first factor will be the group (experimental and control) and the second factor the time (baseline, after completing the implementation of the intervention with NeuronUp APT and six months after the end of the intervention) and the dependent variables, the scores on the measures used.

ELIGIBILITY:
Inclusion Criteria:

1) Be between 18 and 65 years old at the time of the intervention; 2) enter the Acquired Brain Injury Unit of the Aita Menni hospital with a diagnosis of ABI;3) have been hospitalized in the Aita Menni unit for at least 3 weeks;4) the patient must know how to read and write; 5) obtain a score below the 10th percentile in at least one of the attention tests in the screening phase and 6) not present post traumatic amnesia at the start of the study, in the case of patients with TBI.

Exclusion Criteria:

1) Present severe behavioral alterations; 2) have a previous history of neurological disease, psychiatric disorders, intellectual disability, learning disorders and / or substance abuse; 3) have a diagnosis of aphasia; 4) present a score less than or equal 23 in the Mini-mental State Examination (MMSE) and 5) present severe motor or sensory problems that may limit the performance of the tests and the attention rehabilitation program.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited with ABI, aged between 18 and 65, who attend the Acquired Brain Injury Unit of Aita Menni Hospital (Mondragón-Arrasate); specifically, the investigators will focus on participants whose diagnosis is moderate-severe TBI and participants with a diagnosis of stroke in the last three years.
Sampling Method: Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2019-10-30 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Short attention test (BTA): changes in the measure before the intervention (pre-intervention), after the intervention (post-intervention) and six months after the intervention | Pre-intervention, post-intervention (immediately after the intervention) and six months after post-intervention
  The test is used as a measure of divided attention. It can be used in people between 17 and 82 years, it is of individual application with an approximate duration of 10 minutes.
Trail Making Test (TMT A-B): changes in the measure before the intervention (pre-intervention),after the intervention (post-intervention) and six months after the intervention | Pre-intervention, post-intervention (immediately after the intervention) and six months after post-intervention
  The test is used to evaluate attention, psychomotor speed, cognitive flexibility, visual search and executive functions.
Test of Colors and Words (Stroop Test): changes in the measure before the intervention (pre-intervention),after the intervention (post-intervention) and six months after the intervention | Pre-intervention, post-intervention (immediately after the intervention) and six months after post-intervention
  It provides information on the inhibitory capacity of the subject and its resistance to stimulus interference.
Symbol and digit test (SDMT): changes in the measure before the intervention (pre-intervention),after the intervention (post-intervention) and six months after the intervention | Pre-intervention, post-intervention (immediately after the intervention) and six months after post-intervention
  It is a test that involves the conversion of geometric designs into written and / or spoken numerical responses. The test is applied from 8 years to 78 and can be individually or collectively. Because the test consists of geometric figures and numbers, and these are universal symbols of written language, the SDMT test is relatively free of cultural and idiomatic factors and can be applied in different countries and languages.
PASAT test: changes in the measure before the intervention (pre-intervention),after the intervention (post-intervention) and six months after the intervention | Pre-intervention, post-intervention (immediately after the intervention) and six months after post-intervention
  This test is a measure of cognitive function that evaluates the speed and flexibility of the processing of auditory information, as well as the ability to calculate.
Bells Test: changes in the measure before the intervention (pre-intervention),after the intervention (post-intervention) and six months after the intervention | Pre-intervention, post-intervention (immediately after the intervention) and six months after post-intervention
  The Bells Test is used to detect visual inattention in children and adults and it consists of a 21.5 × 28 cm sheet of paper on which seven lines of 35 distractor figures (e.g., bird, key, apple, mushroom, car) and five target figures (bells) are presented. The target figures are arranged so that five of each appears in seven equal columns on the page
Attention Test D2: changes in the measure before the intervention (pre-intervention),after the intervention (post-intervention) and six months after the intervention | Pre-intervention, post-intervention (immediately after the intervention) and six months after post-intervention
  This test is a cancellation task that evaluates the basic processes of selective attention and mental concentration. This instrument also reflects three components of attentional behavior: the speed or amount of work, the quality of work and the relationship between speed and accuracy of attention.
Minimental State Examination (MMSE): changes in the measure before the intervention (pre-intervention),after the intervention (post-intervention) and six months after the intervention | Pre-intervention, post-intervention (immediately after the intervention) and six months after post-intervention
  MMSE is a short and quantitative measurement that can be used to detect cognitive deficits, to assess its severity at a given time, to follow the course of cognitive changes over time and to evaluate the response to a treatment. Several investigations have shown that the MMSE is a reliable and valid instrument in different patient samples and the general population.The scores of MMSE are 0 to 30. In this study the participants need to have a score major 23 for participate. Because, if the score is less or equal 23 in this test, the participant can have an important cognitive deficits.

SECONDARY OUTCOMES:
Hopkins Verbal Learning Test - Revised (HVLT-R): changes in the measure before the intervention (pre-intervention),after the intervention (post-intervention) and six months after the intervention | Pre-intervention, post-intervention (immediately after the intervention) and six months after post-intervention
  It is one of the most used tests to measure learning and verbal memory in the neuropsychological clinical evaluation. It consists of a list of 12 words extracted from 3 different semantic categories.
Test of the complex figure of Rey: changes in the measure before the intervention (pre-intervention),after the intervention (post-intervention) and six months after the intervention | Pre-intervention, post-intervention (immediately after the intervention) and six months after post-intervention
  It is a very useful instrument to evaluate the perceptual organization and visual memory in people with brain damage, evaluate the ability to organize and plan strategies for problem solving, as well as the viso-constructive capacity.
Modified test of classification of Wisconsin cards (M-WCST): changes in the measure before the intervention (pre-intervention),after the intervention (post-intervention) and six months after the intervention | Pre-intervention, post-intervention (immediately after the intervention) and six months after post-intervention
  It is a variation of the Wisconsin Card Classification test created to assess abstract reasoning and the ability to adapt cognitive strategies to the changing environment. It is an individual application test for adults between 18 and 90 years and between the administration time and score add approximately 12 minutes.
Boston Denomination Test (BNT): changes in the measure before the intervention (pre-intervention),after the intervention (post-intervention) and six months after the intervention | Pre-intervention, post-intervention (immediately after the intervention) and six months after post-intervention
  The test consists of naming 60 sheets presented in order of difficulty. Its test-retest reliability coefficients are above 0.77 and has demonstrated good internal consistency with indexes greater than 0, 78.
Phonological and Semantic Verbal Fluency Test: changes in the measure before the intervention (pre-intervention),after the intervention (post-intervention) and six months after the intervention | Pre-intervention, post-intervention (immediately after the intervention) and six months after post-intervention
  These types of tests are highly sensitive to brain damage, so they are commonly administered to people with neurological damage (TBI, multiple sclerosis, dementias, etc.).These tests require the person to be flexible, organize the information and exercise inhibition when necessary.
European Brain Injury Questionnaire (EBIQ): changes in the measure before the intervention (pre-intervention),after the intervention (post-intervention) and six months after the intervention | Pre-intervention, post-intervention (immediately after the intervention) and six months after post-intervention
  It is a self-report that gives us a relative measure of the subjective experience of the cognitive, emotional and social difficulties experienced by people with ABI.
Questionnaire of attention problems: changes in the measure before the intervention (pre-intervention),after the intervention (post-intervention) and six months after the intervention | Pre-intervention, post-intervention (immediately after the intervention) and six months after post-intervention
  This is a questionnaire prepared by the department's research team for this project with the objective of obtaining a measure of how attention problems affect the activities of the patient's daily life, said questionnaire consists of 7 questions, one of them multiple choice.
Moss Attention Rating Scale (MARS): changes in the measure before the intervention (pre-intervention),after the intervention (post-intervention) and six months after the intervention | Pre-intervention, post-intervention (immediately after the intervention) and six months after post-intervention
  It is made up of 22 items, through which an observational rating of the behaviors related to care is obtained. It is useful in evaluations of people with TBI (moderate - severe).
Patient Health Questionnaire (PHQ-9): changes in the measure before the intervention (pre-intervention),after the intervention (post-intervention) and six months after the intervention | Pre-intervention, post-intervention (immediately after the intervention) and six months after post-intervention
  This is a 9-item questionnaire that evaluates the presence of major depressive disorder based on the criteria of the diagnostic and statistical manual of mental disorders (DSM-IV-R). Difference between other depressive symptoms, positive depressive symptoms and negative depressive symptoms.
Generalized Anxiety Disorders Scale (GAD-7): changes in the measure before the intervention (pre-intervention),after the intervention (post-intervention) and six months after the intervention | Pre-intervention, post-intervention (immediately after the intervention) and six months after post-intervention
  This is a 7-item scale that evaluates the presence of generalized anxiety disorder based on the criteria of the diagnostic and statistical manual of mental disorders (DSM-IV-R). The scale has been adapted to Spanish.
Quality of life scale (SF-36): changes in the measure before the intervention (pre-intervention),after the intervention (post-intervention) and six months after the intervention | Pre-intervention, post-intervention (immediately after the intervention) and six months after post-intervention
  consists of 36 questions through which the quality of life related to physical and emotional health, the interference of physical and emotional problems in social life is evaluated, the degree of vitality, energy or fatigue and the general perception of health.
Life Satisfaction Scale (SWLS): changes in the measure before the intervention (pre-intervention),after the intervention (post-intervention) and six months after the intervention | Pre-intervention, post-intervention (immediately after the intervention) and six months after post-intervention
  It is a global measure of satisfaction with life that consists of 5 items. Different studies have used this scale for the evaluation of life satisfaction of people with TBI.
Disability Rating Scale (DRS): changes in the measure before the intervention (pre-intervention),after the intervention (post-intervention) and six months after the intervention | Pre-intervention, post-intervention (immediately after the intervention) and six months after post-intervention
  It is an instrument that evaluates functional recovery in patients with moderate and severe traumatic brain injuries from coma to their return to society, taking into account cognitive function.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Carlos Arango Lasprilla, Principal Investigator — Ikerbasque - Basque Foundation for Science
Locations (1):
- Hospital Aita Menni, Arrasate / Mondragón, Guipúzcoa, Spain

IPD SHARING:
Plan to Share IPD: No
No this data wont be available to other researchers

REFERENCES:
- [Background] Arango-Lasprilla, J., Olabarrieta-Landa, L., Laseca-Zaballa, G., Castrillón -Carvajal, J., & Usuga - Ramos, D. (2019).Traumatic Brain Injury in adults. In Brain damage (pp. 151-201). Mexico D.F: Modern Manual.
- [Background] Areny-Balagueró, M., García-Molina, A., Roig-Rovira, T., Tormos, J., & Jodar-Vicente, M. (2016). Relationship between sensation seeking and patient decision making with harm Acquired brain. Psychology: Advances of Discipline, 10 (1), 25-33.
- [Background] Bate AJ, Mathias JL, Crawford JR. Performance on the Test of Everyday Attention and standard tests of attention following severe traumatic brain injury. Clin Neuropsychol. 2001 Aug;15(3):405-22. doi: 10.1076/clin.15.3.405.10279. PMID 11778779
- [Background] Carvajal Castrillón, J., & Restrepo Pelaez, A. (2013). Theoretical foundations and intervention strategies in neuropsychological rehabilitation in adults with acquired brain damage. CES Psychology Magazine, 6 (2), 135-148.
- [Background] Cermak SA, Katz N, McGuire E, Greenbaum S, Peralta C, Maser-Flanagan V. Performance of Americans and israelis with cerebrovascular accident on the Loewenstein Occupational Therapy Cognitive Assessment (LOTCA). Am J Occup Ther. 1995 Jun;49(6):500-6. doi: 10.5014/ajot.49.6.500. PMID 7645662
- [Background] Cicerone KD. Remediation of "working attention" in mild traumatic brain injury. Brain Inj. 2002 Mar;16(3):185-95. doi: 10.1080/02699050110103959. PMID 11874612
- [Background] de Norena D, Rios-Lago M, Bombin-Gonzalez I, Sanchez-Cubillo I, Garcia-Molina A, Tirapu-Ustarroz J. [Effectiveness of neuropsychological rehabilitation in acquired brain injury (I): attention, processing speed, memory and language]. Rev Neurol. 2010 Dec 1;51(11):687-98. Spanish. PMID 21108231
- [Background] Fish J, Manly T, Emslie H, Evans JJ, Wilson BA. Compensatory strategies for acquired disorders of memory and planning: differential effects of a paging system for patients with brain injury of traumatic versus cerebrovascular aetiology. J Neurol Neurosurg Psychiatry. 2008 Aug;79(8):930-5. doi: 10.1136/jnnp.2007.125203. Epub 2007 Nov 26. PMID 18039889
- [Background] Galbiati S, Recla M, Pastore V, Liscio M, Bardoni A, Castelli E, Strazzer S. Attention remediation following traumatic brain injury in childhood and adolescence. Neuropsychology. 2009 Jan;23(1):40-9. doi: 10.1037/a0013409. PMID 19210031
- [Background] García-Molina, A., Gómez, A., Rodríguez, P., Sánchez-Carrión, R., Zumarraga, L., Enseñat, A., ... Roig-Rovira, T. (2010). Clinical program of cognitive telerehabilitation in craniocerebral trauma. Trauma Fund MAPFRE, 21 (1), 58-63.
- [Background] Greenwald BD, Kapoor N, Singh AD. Visual impairments in the first year after traumatic brain injury. Brain Inj. 2012;26(11):1338-59. doi: 10.3109/02699052.2012.706356. Epub 2012 Aug 16. PMID 22897509
- [Background] Heilman, K., & Valenstein, E. (1993). Clinical Neuropsychology (3rd ed.). New York: Oxford University Press.
- [Background] Ison, M. (2011). Intervention program to improve the attention capacities in Argentine schoolchildren. International Journal of Psychological Research, 4 (2), 72-79.
- [Background] Khan F, Baguley IJ, Cameron ID. 4: Rehabilitation after traumatic brain injury. Med J Aust. 2003 Mar 17;178(6):290-5. doi: 10.5694/j.1326-5377.2003.tb05199.x. PMID 12633489
- [Background] Madigan NK, DeLuca J, Diamond BJ, Tramontano G, Averill A. Speed of information processing in traumatic brain injury: modality-specific factors. J Head Trauma Rehabil. 2000 Jun;15(3):943-56. doi: 10.1097/00001199-200006000-00007. PMID 10785624
- [Background] Marsh NV, Ludbrook MR, Gaffaney LC. Cognitive functioning following traumatic brain injury: A five-year follow-up. NeuroRehabilitation. 2016;38(1):71-8. doi: 10.3233/NRE-151297. PMID 26889800
- [Background] Morton MV, Wehman P. Psychosocial and emotional sequelae of individuals with traumatic brain injury: a literature review and recommendations. Brain Inj. 1995 Jan;9(1):81-92. doi: 10.3109/02699059509004574. PMID 7874099
- [Background] Navarro-Main B, Castano-Leon AM, Munarriz PM, Gomez PA, Rios-Lago M, Lagares A. [Brain injury knowledge in family members of neurosurgical patients]. Neurocirugia (Engl Ed). 2018 Jan-Feb;29(1):1-8. doi: 10.1016/j.neucir.2017.09.007. Epub 2017 Nov 8. Spanish. PMID 29128284
- [Background] Palmese CA, Raskin SA. The rehabilitation of attention in individuals with mild traumatic brain injury, using the APT-II programme. Brain Inj. 2000 Jun;14(6):535-48. doi: 10.1080/026990500120448. PMID 10887887
- [Background] Parasuraman R, Mutter SA, Molloy R. Sustained attention following mild closed-head injury. J Clin Exp Neuropsychol. 1991 Sep;13(5):789-811. doi: 10.1080/01688639108401090. PMID 1955532
- [Background] Quedaza, M. (2011). Acquired Brain Damage (DCA) in Spain: main results from the AGE-2008 Survey. Bulletin of the State Disability Observatory, 3, 39-59.
- [Background] Rios-Lago M, Munoz-Cespedes JM, Paul-Lapedriza N. [Attentional impairment after traumatic brain injury: assessment and rehabilitation]. Rev Neurol. 2007 Mar 1-15;44(5):291-7. Spanish. PMID 17342680
- [Background] Sander AM, Seel RT, Kreutzer JS, Hall KM, High WM Jr, Rosenthal M. Agreement between persons with traumatic brain injury and their relatives regarding psychosocial outcome using the Community Integration Questionnaire. Arch Phys Med Rehabil. 1997 Apr;78(4):353-7. doi: 10.1016/s0003-9993(97)90225-2. PMID 9111453
- [Background] Sohlberg, M. M, Johnson, L., Paule, L., Raskin, S. A., & Mateer, C. A. (2001). Attention process training-II: A program to address attentional deficits for persons with mild cognitive dysfunction (2nd ed.). Wake Forest: NC: Lash & Associates
- [Background] Sohlberg MM, Mateer CA. Effectiveness of an attention-training program. J Clin Exp Neuropsychol. 1987 Apr;9(2):117-30. doi: 10.1080/01688638708405352. PMID 3558744
- [Background] Sohlberg MM, McLaughlin KA, Pavese A, Heidrich A, Posner MI. Evaluation of attention process training and brain injury education in persons with acquired brain injury. J Clin Exp Neuropsychol. 2000 Oct;22(5):656-76. doi: 10.1076/1380-3395(200010)22:5;1-9;FT656. PMID 11094401
- [Background] Varas-Arias MT, Rodriguez-Palero S. [Rehabilitation treatment in child and youth patients with acquired brain injury]. Rev Neurol. 2017 May 17;64(s03):S1-S7. Spanish. PMID 28524211
- [Background] Wassenberg R, Max JE, Lindgren SD, Schatz A. Sustained attention in children and adolescents after traumatic brain injury: relation to severity of injury, adaptive functioning, ADHD and social background. Brain Inj. 2004 Aug;18(8):751-64. doi: 10.1080/02699050410001671775. PMID 15204316
- [Background] Whyte J, Hart T, Ellis CA, Chervoneva I. The Moss Attention Rating Scale for traumatic brain injury: further explorations of reliability and sensitivity to change. Arch Phys Med Rehabil. 2008 May;89(5):966-73. doi: 10.1016/j.apmr.2007.12.031. PMID 18452747
- [Background] Wilson, B. A. (2013). Neuropsychological rehabilitation: State of the science. South African Journal of Psychology, 43(3), 267-277.
- [Background] Yeates KO, Armstrong K, Janusz J, Taylor HG, Wade S, Stancin T, Drotar D. Long-term attention problems in children with traumatic brain injury. J Am Acad Child Adolesc Psychiatry. 2005 Jun;44(6):574-84. doi: 10.1097/01.chi.0000159947.50523.64. PMID 15908840

DOCUMENTS (2):
  • Study Protocol (2021-02-12): https://cdn.clinicaltrials.gov/large-docs/14/NCT04214314/Prot_004.pdf
  • Informed Consent Form (2021-02-12): https://cdn.clinicaltrials.gov/large-docs/14/NCT04214314/ICF_005.pdf